CLINICAL TRIAL: NCT01827956
Title: Role of FCγRIIIA and FCγRIIA Receptor Polymorphisms in Cetuximab Activity Used in Palliative Treatment of Upper Aerodigestive Tract Tumours
Brief Title: Role of FCγRIIIA and FCγRIIA Receptor Polymorphisms
Acronym: FCR-VADS
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB2009-24
Record Dates: First submitted 2012-11-05; First posted 2013-04-10 (Estimated); Results first posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Upper Gingival Squamous Cell Carcinoma
Keywords: Upper aero-digestive tract tumours; FCGR3A and FCGR2A receptor polymorphism; Cetuximab efficacy
MeSH Terms: interventions — Cetuximab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UGSCS: Patients with Upper Gingival Squamous Cell Carcinoma initiating Cetuximab treatment
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Blood sample for identifying the polymorphism of FCGR3A and FCGR2A genes

SUMMARY:
Hypothesis:

Cetuximab, an anti-EGFR antibody, is used with radiotherapy in the treatment of locally advanced and inoperable upper aerodigestive tract cancers. Actually, no predictive biomarkers of Cetuximab antitumor activity are known in this setting. It has been shown recently that FCγRIIIA and FCγRIIA receptor polymorphisms played a role in antitumor activity of trastuzumab and cetuximab.

The investigators therefore hypothesized that FCγRIIIA and FCγRIIA receptor polymorphisms may play a predictive role in Cetuximab effectiveness in upper aerodigestive tract cancers with recurrence or metastatic disease that make them inaccessible to loco regional treatment.

DETAILED DESCRIPTION:
Hypothesis:

Cetuximab, an anti-EGFR antibody, is used with radiotherapy in the treatment of locally advanced and inoperable upper aerodigestive tract cancers. Actually, no predictive biomarkers of Cetuximab antitumor activity are known in this setting. It has been shown recently that FCγRIIIA and FCγRIIA receptor polymorphisms played a role in antitumor activity of trastuzumab and cetuximab.

We therefore hypothesized that FCγRIIIA and FCγRIIA receptor polymorphisms may play a predictive role in Cetuximab effectiveness in upper aerodigestive tract cancers with recurrence or metastatic disease that make them inaccessible to loco regional treatment.

This study is a multicentre prospective pharmacogenetic observational study, conducted on locally advanced and inoperable upper aerodigestive tract cancers.

* Blood sample for polymorphism identification (5 ml plastic tube with EDTA, taken at the start of treatment, at the same time as the blood samples routinely taken as part of standard care)
* Collection of medical data at inclusion and at 4 months

ELIGIBILITY:
Inclusion Criteria:

* Patient with recurrent or metastatic squamous cell carcinomas of the upper aero-digestive tract
* Patient with loco-regional extension not readily treatable
* 18 years
* Follow up in participant center
* Patient information and consent for study participation
* Patient presented in multidisciplinary meeting (RCP) in Aquitaine and for whom a treatment containing cetuximab has been proposed
* Belong to a social security system

Exclusion Criteria:

* Pregnancy
* Patient with psychological, social, family or geographical reason, who could not be treated or monitored regularly by study criteria,
* Patients deprived of liberty or under guardianship or who could not give consent for study participation
* Inclusion in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Squamous cell carcinomas of the upper aero-digestive tract recurrent or metastatic.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ROBERT Jacques, PU-PH, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UGSCS
Started | 121
Completed | 118
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | UGSCS
Number analyzed (Participants) | 121
Age, Continuous [Median (Full Range); unit: years] | 60.9 [30.6 to 81.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 96
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 121

OUTCOME MEASURES:

1. Primary Outcome: Polymorphism of FCGR2 Gene
Description: Polymorphism of FCGR2A gene is expressed according to 3 modalities : RR / RH / HH
  Genomic DNA will be extracted from whole blood tubes and redissolved in 100 µl 1× TE buffer and purified on GFX columns (Amersham-Biosciences). The quantity and quality of the DNA will be checked by agarose gel electrophoresis in the presence of ethidium bromide. Polymorphisms will be detected by PCR followed by pyrosequencing.
Time Frame: At treatment initiation
Population: Population with FCGR2 gene contributive results
Measure: Count of Participants; unit: Participants
Arm/Group | UGSCS
Number analyzed (Participants) | 118
Participants
  RR | 29
  RH | 53
  HH | 36

2. Primary Outcome: Polymorphism of FCGR3A Gene
Description: Polymorphism of FCGR3A gene is expressed according to 3 modalities : FF / FV / VV.
  Genomic DNA will be extracted from whole blood tubes and redissolved in 100 µl 1× TE buffer and purified on GFX columns (Amersham-Biosciences). The quantity and quality of the DNA will be checked by agarose gel electrophoresis in the presence of ethidium bromide. Polymorphisms will be detected by PCR followed by pyrosequencing.
Time Frame: At treatment initiation
Population: Population with FCGR3 gene contributive results
Measure: Count of Participants; unit: Participants
Arm/Group | UGSCS
Number analyzed (Participants) | 117
Participants
  FF | 54
  FV | 48
  HH | 15

3. Secondary Outcome: 4-month Non-progression Rate According to the Polymorphism
Description: The primary endpoint is the 4-month non-progression rate assessed according to RECIST criteria (or according to a clinical assessment if the patient does not undergo radiological examination). The response will be considered "no progression" in the following cases: complete response, partial response, or stable disease. In other cases (disease progression or unevaluable), the disease will be considered to be progressing.
  Response will be assessed at enrollment and at 4 months or until the first of the following events: disease progression or patient death.
Time Frame: 4 months after treatment initiation
Population: Population with either FCGR2 gene contributive results or FCGR3 gene contributive results
Measure: Count of Participants; unit: Participants
Groups:
- UGSCS With Polymorphism "FCG2RA = HH or FCG3RA = VV"; UGSCS With Polymorphism Other Than "FCG2RA = HH or FCG3RA = VV": Patients with Upper Gingival Squamous Cell Carcinoma initiating Cetuximab treatment
  Cetuximab: Blood sample for identifying the polymorphism of FCGR3A and FCGR2A genes
Arm/Group | UGSCS With Polymorphism "FCG2RA = HH or FCG3RA = VV" | UGSCS With Polymorphism Other Than "FCG2RA = HH or FCG3RA = VV"
Number analyzed (Participants) | 41 | 77
Participants
  Non progression | 18 | 47
  Progression | 23 | 30

4. Secondary Outcome: Overall Survival Rate
Description: Overall survival: defined as the time between the first cycle of chemotherapy and the date of death, all causes. In the absence of death confirmation, survival data are censored from the date of last news
Time Frame: 12 months
Population: Population with either FCGR2 gene contributive results and FCGR3 gene contributive results and follow-up data available
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | UGSCS With Polymorphism "FCG2RA = HH or FCG3RA = VV" | UGSCS With Polymorphism Other Than "FCG2RA = HH or FCG3RA = VV"
Number analyzed (Participants) | 41 | 77
months | 10.16 [6.57 to 15.25] | 10.48 [6.97 to 14.00]

ADVERSE EVENTS:
Time Frame: 24 months
Description: Serious Adverse Events and other NON Serious Adverse Events were not collected
Arm/Group | UGSCS
All-Cause Mortality (participants affected / at risk) | 87/121
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes